CLINICAL TRIAL: NCT00061048
Title: Phase II Study of the Efficacy and Toxicity of Campath-1H in the Therapy of Adult T-Cell Leukemia
Brief Title: Campath-1H for Treating Adult T-Cell Leukemia/Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Thomas A. Waldmann, M.D., National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030194; 03-C-0194 (Other: Clinical Center (CC), National Institutes of Health (NIH)); 030194 (Other: Clinical Center (CC), National Institutes of Health (NIH)); NCT00064155 (obsolete NCT alias)
Record Dates: First submitted 2003-05-20; First posted 2003-05-21 (Estimated); Results first posted 2011-06-08 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Acute T-Cell Leukemia-Lymphoma
Keywords: Monoclonal Antibody; HTLV-1; CD52; Flow Cytometry; Antibody Saturation; Adult T-Cell Leukemia (ATL); ATL
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Campath-1H (Experimental): Infusion of Campath-1H 3 mg on day # 1, 10 mg on day #2, and 30 mg day # 3 followed by maintenance Campath-1H 30 mg intravenously three times per week.
  Interventions: Biological: Alemtuzumab

INTERVENTIONS:
Biological: Alemtuzumab — Infusion of Campath-1H 3 mg on day # 1, 10 mg on day #2, and 30 mg day # 3 followed by maintenance Campath-1H 30 mg intravenously three times per week. Patients are eligible to receive a maximum of 12 weeks of maintenance Campath-1H treatment.

SUMMARY:
This study will examine the safety and effectiveness of Alemtuzumab (Campath-1H) for treating patients with adult T-cell leukemia/lymphoma (ATL). ATL is caused by a virus called human T-cell lymphotrophic virus type-1 (HTLV-1) that infects lymphocytes (white blood cells) called T-cells. Cancerous cells can be found not only in the blood, but also in the skin, lungs, lymph nodes, liver, bone, bone marrow, spleen, and meninges (tissues covering the brain). There are four categories of ATL, based on the aggressiveness of disease-smoldering, chronic, lymphoma, and acute. Campath-1H is a monoclonal antibody that attaches to and kills normal and cancerous lymphocytes, including T cells. Although Campath-1H is an experimental drug for treating ATL, it is approved by the Food and Drug Administration for treating chronic lymphocytic leukemia.

Patients 18 years of age and older with any type of ATL except smoldering may be eligible for this study. Candidates are screened with a medical history and physical examination, photos of skin lesions, measurement of lesions such as lymph nodes and skin nodules, blood and urine tests, electrocardiogram (EKG), chest x-ray, computed tomography (CT) scan or ultrasound of the abdomen, skin biopsy, bone marrow aspirate and biopsy, skin test, and lumbar puncture (spinal tap). Participants undergo treatment in two phases, as follows:

* Dose escalation phase: Patients receive an infusion of Campath-1H daily for three days. The initial dose is low and is increased daily as long as there are no side effects, or only mild reactions, until the patient is receiving the maximum dose of 30 milligrams per day.
* Stable dose phase: Patients receive infusions of Campath-1H 30 mg three times a week for up to 12 weeks.

In addition to treatment, patients are evaluated with the following tests and procedures:

* History and physical examination every 4 weeks.
* Blood tests every 4 weeks.
* CT scans to measure the size of the tumors every 4 weeks.
* Skin biopsies (if skin disease is present) and lymph note aspirates: Up to five biopsies and five aspirates may be taken to help diagnose the disease and evaluate the effect of Campath-1H on the cancer.
* Bone marrow biopsy: This procedure may be done to document or monitor disease progress.

Patients receive treatment for up to 12 weeks. Treatment may stop earlier if the patient achieves a complete response before the end of 12 weeks. Patients completing the study are followed periodically with a history and physical examination, blood and urine tests, tumor evaluation, skin biopsy and skin testing. They are seen monthly at first and then at 3-month intervals the first year; every 4 months the second year, every 6 months for the third through fifth years, and then yearly.

DETAILED DESCRIPTION:
Background:

Adult T-cell leukemia/lymphoma (ATL) is an aggressive lymphoproliferative disorder caused by an infection with the human T-cell lymphotrophic virus type-1 (HTLV-1).

ATL is characterized by rapidly rising peripheral blood leukemia cell counts, lymphadenopathy, lytic bone lesions, hepatosplenomegaly, and skin and solid organ involvement by tumor.

Chemotherapy has shown modest activity and the treatment of ATL has remained largely undefined and the survival of ATL patients poor.

The CD52 surface glycoantigen is overexpressed on ATL cells.

Alemtuzumab (Campath-1H) is a humanized rat monoclonal antibody that binds to CD52 and is cytotoxic.

In preclinical models, Campath-1H inhibited tumor growth and improved the survival of Non-obese diabetic (NOD)/severe combined immune deficiency (SCID) mice injected with human MET-1 ATL cells.

Objectives:

To determine the efficacy of Campath-1H in the treatment of ATL.

To define the time course of Campath-1H saturation in patients with ATL.

To define the toxicity of Campath-1H in patients with ATL.

Eligibility:

Patients with HTLV-I-associated adult T-cell leukemia.

More than 10% of the malignant cells must express CD52 and CD25.

Patients must have measurable disease.

The patient must have a granulocyte count of at least 1000/mm(3) and a platelet count of greater than or equal to 50,000/mm(3).

Design:

A single institution non-randomized open-label Phase II trial.

This trial will recruit a maximum of 30 eligible patients.

Patients will receive antimicrobial and antiviral prophylaxis while on-study due to the known immunosuppressive effects of Campath-1H.

Patients will receive I.V. Campath-1H 3 mg on day 1, 10 mg on day 2, and 30 mg day 3 followed by maintenance Campath-1H 30 mg I.V. three time per week.

Patients will be evaluated for response and continuation of Campath-1H therapy after weeks 4 and 8 of maintenance treatment.

Patients are eligible to receive a maximum of 12 weeks of maintenance Campath-1H treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have serum antibodies directed to Human T-lymphotropic Virus Type 1 (HTLV-1).
* All patients must have a histologically confirmed diagnosis of adult T- cell leukemia/lymphoma and more than 10% of the malignant cells must express CD52 and CD25.
* All stages of Tac-expressing adult T-cell leukemia except smoldering are eligible: patients with chronic, lymphoma or acute Acute T-cell leukemia/lymphoma (ATL) are eligible.
* Patients must have measurable disease. All patients with greater than 10% abnormal (i.e. Tac homogeneous strongly expressing) peripheral blood mononuclear cell (PBMC)in the peripheral blood will be deemed to have measurable disease.
* The patient must have a granulocyte count of at least 100/mm(3) and a platelet count of greater than or equal to 50,000/mm(3).
* Patients must have a creatinine of less than 3.0 mg/dl.
* Omission of cytotoxic chemotherapy for ATL for 3 weeks prior to entry into the trial is required. However patients receiving a stable dose of corticosteroids for at least three to four weeks without evidence of tumor response will be eligible.
* Patients must have a life expectancy of greater than 2 months.
* Eligible patients must be greater than or equal to 18 years old. There is no upper age limit.
* Patients must have serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) value less than or equal to 2.5-fold greater than the upper limit of normal and bilirubin less than or equal to 3.0/dl. If a liver function test is judged to be elevated due to the underlying ATL, this parameter will be considered an unevaluable parameter for toxicity determinations.
* Patients must be able to understand and sign an Informed Consent form.
* All patients must use adequate contraception during participation in this trial and for three months after completing therapy.

Exclusion Criteria:

* Patients with symptomatic leukemic meningitis will be excluded. However patients that have both ATL and another HTLV-1-associated disease, tropical spastic paraparesis (TSP) will be included.
* Pregnant and nursing patients are not eligible for the study. Because the effects of CAMPATH-1H on the developing fetus are unknown pregnant women will be excluded. Breast-feeding in patients with HTLV-1 infection is contraindicated because of the risk of transmission of the virus to the child. In addition, CAMPATH-1H may be present in breast milk and produce adverse events in the breast-feeding child.
* Human immunodeficiency virus (HIV) positive patients are excluded from the study. CAMPATH-1H may produce a different pattern of toxicities in patients with HIV infection and in addition the depletion of T cells produced by CAMPATH-1H may have adverse effects on HIV positive individuals.
* Patients with smoldering ATL are excluded.
* Patients with previously received Campath-1GH are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2003-05; Primary Completion 2009-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Waldmann, M.D., Principal Investigator — NCI, NIH
Locations (1):
- National Institutes of Health, National Cancer Institute, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kohler G, Milstein C. Continuous cultures of fused cells secreting antibody of predefined specificity. 1975. Biotechnology. 1992;24:524-6. No abstract available. PMID 1422065
- [Background] Catane R, Longo DL. Monoclonal antibodies for cancer therapy. Isr J Med Sci. 1988 Sep-Oct;24(9-10):471-6. PMID 3060441
- [Background] Dickman S. Antibodies stage a comeback in cancer treatment. Science. 1998 May 22;280(5367):1196-7. doi: 10.1126/science.280.5367.1196. No abstract available. PMID 9634400
- [Derived] Chen J, Pise-Masison CA, Shih JH, Morris JC, Janik JE, Conlon KC, Keating A, Waldmann TA. Markedly additive antitumor activity with the combination of a selective survivin suppressant YM155 and alemtuzumab in adult T-cell leukemia. Blood. 2013 Mar 14;121(11):2029-37. doi: 10.1182/blood-2012-05-427773. Epub 2013 Jan 15. PMID 23321252
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information Portal — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas — http://jco.ascopubs.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Anticipate enrolling 10-12 patients per year into the Campath-1H trial. Thus, if the trial goes to completion (2nd stage)we anticipate enrolling the 29 patients in approximately 2.5 years.
Groups:
- Campath-1H Treatment of Adult T-cell Leukemia (ATL): Intravenous Campath-1H 3 mg on day #1, 10mg on day #2, and 30mg on day #3 followed by maintenance Campath-1H 30 mg intravenously three times per week. Patients are eligible to receive a maximum of 12 weeks of maintenance Campath-1H treatment.
Period: Overall Study
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Started | 29
Completed | 7 (Began protocol specified follow-up period.)
Not Completed | 22
Not completed — Adverse Event | 2
Not completed — disease progression | 20

BASELINE CHARACTERISTICS:
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 52.54 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants with response and utilizes the International Standardized workshop definition.
  Complete response(CR)-Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related symptoms if present before therapy and normalization of those biochemical abnormalities (for example LDH) definitely assignable to the lymphoma.
  Please see the protocol Link module for the full criteria if desired.
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Number analyzed (Participants) | 29
percentage of participants | 52 [32.5 to 70.6]

2. Primary Outcome: Overall Survival
Description: Time between the first day of treatment to the day of death.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Number analyzed (Participants) | 29
months | 5.9 [4.7 to 8.7]

3. Primary Outcome: Time to Progression
Description: Time between the first day of treatment to the day of disease progression which is defined as a persistent (at least two determinations) doubling of the peripheral blood leukemic cell count, the development of new lesions, or Ca elevations that are uncontrolled by conventional therapeutic procedures.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Number analyzed (Participants) | 29
months | 2.0 [1.0 to 3.9]

4. Secondary Outcome: Cell Surface Expression of CD52 on Tumor Cells
Description: The CD52 antibody-binding capacity (ABC) value is the measurement of the mean value of the maximum capacity of each cell to bind the anti-CD52 and when determined under conditions of saturating levels of antibody measures number of mean surface CD52 antigens per cell. CD52 ABC is negative when 100% saturation by therapeutic antibody is achieved.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ABC value
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Number analyzed (Participants) | 29
ABC value | 82.15 (13.7)

5. Secondary Outcome: The Number of Participants With Adverse Events
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Number analyzed (Participants) | 29
participants | 8

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Campath-1H Treatment of Adult T-cell Leukemia (ATL)
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath-1H Treatment of Adult T-cell Leukemia (ATL) (N=29)
CARDIOVASCULAR (GENERAL):: Hypotension (Vascular disorders) | 1 (1) — cardiovascular; orthostatic hypotension
CONSTITUTIONAL SYMPTOMS:: Constitutional Symptoms-Other (death) (General disorders) | 2 (2)
CONSTITUTIONAL SYMPTOMS:: Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
CONSTITUTIONAL SYMPTOMS:: Rigors, chills (General disorders) | 1 (1) — Infusional reaction
ENDOCRINE:: Endocrine-Other (Endocrine:hyperthyroidism graves disease) (Endocrine disorders) | 1 (1)
GASTROINTESTINAL:: Vomiting (Gastrointestinal disorders) | 1 (1) — Infusional reaction
INFECTION/FEBRILE NEUTROPENIA:: Infection without neutropenia (Infections and infestations) | 1 (1) — Infection: strongyloidosis
METABOLIC/LABORATORY:: Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
NEUROLOGY:: Neurology-Other (Unresponsiveness) (Nervous system disorders) | 1 (1)
OCULAR/VISUAL:: Vision-blurred vision (Eye disorders) | 1 (1) — Blurred vision due to uveitis
PULMONARY:: Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY:: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath-1H Treatment of Adult T-cell Leukemia (ATL) (N=29)
ALLERGY/IMMUNOLOGY:: Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2) — Allergy: infusional reaction
ALLERGY/IMMUNOLOGY:: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
BLOOD/BONE MARROW:: Hemoglobin (Investigations) | 20 (81) — Anemia Hemoglobin
BLOOD/BONE MARROW:: Leukocytes (total WBC) (Investigations) | 15 (106) — Decrease WBC
BLOOD/BONE MARROW:: Lymphopenia (Investigations) | 18 (26) — Lymphopenia Low lymphocytes
BLOOD/BONE MARROW:: Neutrophils/granulocytes (ANC/AGC) (Investigations) | 11 (54) — ANC
BLOOD/BONE MARROW:: Platelets (Investigations) | 16 (41) — Platelets
CARDIOVASCULAR (ARRHYTHMIA):: Cardiovascular/Arrhythmia-Other (irregular heartbeat)) (Cardiac disorders) | 1 (1)
CARDIOVASCULAR (ARRHYTHMIA):: Sinus bradycardia (Cardiac disorders) | 1 (2) — Sinus bradycardia
CARDIOVASCULAR (ARRHYTHMIA):: Sinus tachycardia (Cardiac disorders) | 5 (13) — Sinus tachycardia
CARDIOVASCULAR (ARRHYTHMIA):: Vasovagal episode (Cardiac disorders) | 3 (3) — Vasovagal episode, Fall
CARDIOVASCULAR (GENERAL):: Edema (Cardiac disorders) | 5 (7) — Bilat foot, legs, ankle edema Edema: face, forearm, hands, legs Facial swelling Ankles to knees edema Pitting
CARDIOVASCULAR (GENERAL):: Hypertension (Vascular disorders) | 2 (2) — Hypertension
CARDIOVASCULAR (GENERAL):: Hypotension (Vascular disorders) | 11 (15) — Hypotension Orthostatic hypotension only after Campath infusions
CARDIOVASCULAR (GENERAL):: Phlebitis (superficial) (Cardiac disorders) | 2 (2)
COAGULATION:: Partial thromboplastin time (PTT) (Investigations) | 4 (5)
COAGULATION:: Prothrombin time (PT) (Investigations) | 2 (2)
CONSTITUTIONAL SYMPTOMS:: Fatigue (lethargy, malaise, asthenia) (General disorders) | 5 (6) — Fatigue Fatigue (lethargy, malaise, asthenia) Fever
CONSTITUTIONAL SYMPTOMS:: Fever (in the absence of neutropenia, where neutropenia is defined as AGC< (General disorders) | 22 (68) — Fever Infusional reaction
CONSTITUTIONAL SYMPTOMS:: Rigors, chills (General disorders) | 25 (48) — Chills Infusional reaction Mild chills Rigors Rigors, chills Chills with Campath Infusional reaction occurred overnight
CONSTITUTIONAL SYMPTOMS:: Sweating (diaphoresis) (General disorders) | 1 (1) — Sweating (diaphoresis)
CONSTITUTIONAL SYMPTOMS:: Weight gain (General disorders) | 1 (1) — Ankle edema (increase wt)
CONSTITUTIONAL SYMPTOMS:: Weight loss (General disorders) | 3 (6) — Weight loss
DERMATOLOGY/SKIN:: Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (2) — Abdominal bruising, ecchymosis
DERMATOLOGY/SKIN:: Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
DERMATOLOGY/SKIN:: Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) — Derm: swelling in right arm injection site reaction
DERMATOLOGY/SKIN:: Pruritus (Skin and subcutaneous tissue disorders) | 8 (10) — Itching
DERMATOLOGY/SKIN:: Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 (12) — Skin rash papules (on breast, chest)
DERMATOLOGY/SKIN:: Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 11 (15) — Derm: hives, infusion reaction 20 min post Campath On thighs and stomach
ENDOCRINE:: Hypothyroidism (Endocrine disorders) | 1 (2)
GASTROINTESTINAL:: Anorexia (Gastrointestinal disorders) | 6 (6)
GASTROINTESTINAL:: Constipation (Gastrointestinal disorders) | 9 (13)
GASTROINTESTINAL:: Diarrhea patients without colostomy (Gastrointestinal disorders) | 10 (11)
GASTROINTESTINAL:: Dyspepsia/heartburn (Gastrointestinal disorders) | 3 (3)
GASTROINTESTINAL:: Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Flatulence (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal-Other (Abdominal distention) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Mouth dryness (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL:: Nausea (Gastrointestinal disorders) | 11 (13) — Infusional reaction
GASTROINTESTINAL:: Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 3 (5) — Tongue and oral mucosa stomatitis
GASTROINTESTINAL:: Vomiting (Gastrointestinal disorders) | 10 (12) — Infusional reaction
HEMORRHAGE:: Epistaxis (Blood and lymphatic system disorders) | 7 (7) — Dry due to membrane inflammation
HEMORRHAGE:: Vaginal bleeding (Blood and lymphatic system disorders) | 1 (1) — Spotting
HEPATIC:: Alkaline phosphatase (Hepatobiliary disorders) | 8 (10)
HEPATIC:: Bilirubin (Hepatobiliary disorders) | 5 (11)
HEPATIC:: GGT (Gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 1 (1)
HEPATIC:: Hypoalbuminemia (Hepatobiliary disorders) | 14 (38)
HEPATIC:: SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 12 (22) — Aspartate aminotransferase
HEPATIC:: SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 9 (14) — Alanine aminotransferase
INFECTION/FEBRILE NEUTROPENIA:: Catheter-related infection (Blood and lymphatic system disorders) | 1 (1)
INFECTION/FEBRILE NEUTROPENIA:: Febrile neutropenia (fever of unknown origin without clinically or m (Blood and lymphatic system disorders) | 1 (1) — Fever
INFECTION/FEBRILE NEUTROPENIA:: Infection (documented clinically or microbiologically) with grade 3 (Blood and lymphatic system disorders) | 1 (1)
INFECTION/FEBRILE NEUTROPENIA:: Infection without neutropenia (Blood and lymphatic system disorders) | 9 (17) — CMV CMV(+) Methicillin staphyloccocus aureus (+) Nares (-) Sinus infection (staph aureus) Infection without neutropenia streptococcus Infection: strongyloidosis Left inguinal cellulitis-redness
INFECTION/FEBRILE NEUTROPENIA:: Infection/Febrile Neutropenia-Other (CMV antigenemia) (Blood and lymphatic system disorders) | 5 (5)
LYMPHATICS:: Lymphatics (Blood and lymphatic system disorders) | 1 (1) — Left inguinal swelling
LYMPHATICS:: Lymphatics-Other (Lymphocytes) (Blood and lymphatic system disorders) | 1 (1)
METABOLIC/LABORATORY:: Amylase (Investigations) | 2 (3) — Amylase
METABOLIC/LABORATORY:: Bicarbonate (Investigations) | 2 (2) — Bicarbonate
METABOLIC/LABORATORY:: CPK (creatine phosphokinase) (Investigations) | 2 (2)
METABOLIC/LABORATORY:: Hypercalcemia (Investigations) | 5 (14) — Hypercalcemia
METABOLIC/LABORATORY:: Hypercholesterolemia (Investigations) | 1 (1) — Hypercholesterolemia
METABOLIC/LABORATORY:: Hyperglycemia (Investigations) | 13 (34) — Hyperglycemia
METABOLIC/LABORATORY:: Hyperkalemia (Investigations) | 1 (3)
METABOLIC/LABORATORY:: Hypermagnesemia (Investigations) | 7 (12) — Hypermagnesemia
METABOLIC/LABORATORY:: Hypernatremia (Investigations) | 1 (1) — Hypernatremia
METABOLIC/LABORATORY:: Hyperuricemia (Investigations) | 6 (12) — Hyperuricemia
METABOLIC/LABORATORY:: Hypocalcemia (Investigations) | 5 (20) — Hypocalcemia
METABOLIC/LABORATORY:: Hypoglycemia (Investigations) | 4 (4) — Hypoglycemia
METABOLIC/LABORATORY:: Hypokalemia (Investigations) | 9 (18) — Hypokalemia
METABOLIC/LABORATORY:: Hypomagnesemia (Investigations) | 9 (33) — Hypomagnesemia
METABOLIC/LABORATORY:: Hyponatremia (Investigations) | 10 (27) — Hyponatremia
METABOLIC/LABORATORY:: Hypophosphatemia (Investigations) | 6 (19) — Hypophosphatemia
METABOLIC/LABORATORY:: Lipase (Investigations) | 1 (1)
METABOLIC/LABORATORY:: Metabolic/Laboratory-Other (Lactate) (Investigations) | 1 (1)
NEUROLOGY:: Dizziness/lightheadedness (Nervous system disorders) | 4 (4)
NEUROLOGY:: Insomnia (Psychiatric disorders) | 5 (5)
NEUROLOGY:: Mood alteration-anxiety, agitation (Psychiatric disorders) | 1 (1)
NEUROLOGY:: Mood alteration-depression (Psychiatric disorders) | 1 (1)
NEUROLOGY:: Neuropathy - cranial (Nervous system disorders) | 1 (1)
NEUROLOGY:: Neuropathy - motor (Nervous system disorders) | 3 (3) — Tremor
OCULAR/VISUAL:: Dry eye (Eye disorders) | 1 (1)
OCULAR/VISUAL:: Ocular/Visual-Other (Ocular other: uveitis) (Eye disorders) | 1 (1)
OCULAR/VISUAL:: Tearing (watery eyes) (Eye disorders) | 1 (1)
OCULAR/VISUAL:: Vision-blurred vision (Gastrointestinal disorders) | 2 (2)
OCULAR/VISUAL:: Vision-double vision (diplopia) (Eye disorders) | 2 (2)
OCULAR/VISUAL:: Vision-photophobia (Eye disorders) | 1 (1)
PAIN:: Abdominal pain or cramping (Gastrointestinal disorders) | 2 (2)
PAIN:: Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN:: Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) — During infusion, probable bone marrow involvement with disease
PAIN:: Chest pain (non-cardiac and non-pleuritic) (General disorders) | 4 (4)
PAIN:: Earache (otalgia) (Ear and labyrinth disorders) | 1 (1)
PAIN:: Headache (Nervous system disorders) | 7 (11)
PAIN:: Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 7 (13) — Back pain Generalized achiness/pain Low back pain Low back, hip pain Right thoracic pain muscular Tendonitis right shoulder Back abdominal pain
PAIN:: Pain-Other (Dental-anterior pillars tender;Foot, sharp and intermittent;Right eye ache) (Nervous system disorders) | 6 (7) — Peripherally inserted central catheter site pain Pain other: pain in eyes Pain: in right finger Pain: in right shoulder
PAIN:: Pelvic pain (Reproductive system and breast disorders) | 1 (1) — Left inguinal pain
PAIN:: Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Pain: right inguinal, (new lymph node)
PULMONARY:: Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
PULMONARY:: Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PULMONARY:: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (5) — Infusional reaction Infusional reaction, occurred overnight
PULMONARY:: Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY:: Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RENAL/GENITOURINARY:: Creatinine (Renal and urinary disorders) | 3 (5) — Creatinine
RENAL/GENITOURINARY:: Hemoglobinuria (Renal and urinary disorders) | 1 (1)
RENAL/GENITOURINARY:: Proteinuria (Renal and urinary disorders) | 3 (4) — Proteinuria
RENAL/GENITOURINARY:: Renal/Genitourinary-Other (Urine positive for white blood cells) (Renal and urinary disorders) | 2 (2) — UTI
DERMATOLOGY/SKIN::Dermatology/Skin-Other(Thumb swelling) (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No